CLINICAL TRIAL: NCT05541094
Title: Impact of Vitamin D Fortification of Milk and Oil on Serum Vitamin D Concentrations - An Effectiveness Study
Brief Title: Study of Vitamin D Fortification of Milk and Oil
Acronym: Tata
Status: Completed | Type: Observational
Sponsor: Dr. Anuradha Khadilkar (Other)
Collaborators: TATA Trusts (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Anuradha Khadilkar, Deputy Director at HCJMRI Pune, Hirabai Cowasji Jehangir Medical Research Institute
Organization: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Other Study IDs: TVDFT
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fortified Arm: Individuals from families who are consume fortified milk + oil
- Unfortified Arm: families habitually consuming unfortified milk and oil

SUMMARY:
It is a two-year longitudinal effectiveness study. A comparative study with a case-control design. Study will be conducted in Pune city. A total of up to 100 families (50 families per group) will be recruited. The test group will consist of families consuming fortified milk and oil and the control group will consist of families consuming non fortified milk and oil. Individuals between the age 5-18 years, 18-50 years and more than 50 years will be enrolled. Families which intend to stay in the city for the next 2 years, willing to continue with the same brand of milk and oil for the next 2 years, children living with their biological parents and families willing to sign consent form, will be enrolled in the study. Individuals having chronic illnesses likely to affect vitamin D concentrations and those allergic to milk will be excluded.

DETAILED DESCRIPTION:
Study design: A two-year longitudinal effectiveness study Sample selection: Hundred families will be selected for this study, 50 in each group.

For the test group, people/families buying the standardized milk habitually will be identified and offered the study, an ethics approval would be obtained before commencing the study. After a consent is signed, a home visit will be made and family will be given information about the study.

Individuals from families who consume standardized fortified milk + fortified oil will be offered the study. The control group will consist of families consuming unfortified milk and oil. Thus, families habitually consuming unfortified milk and oil (from 'ghanas') will be offered the study.

ELIGIBILITY:
Inclusion Criteria: Age between 5 to 80 years at the time of enrolment, Intention to stay in the city for the next two years, Families willing to continue with same brand of oil and milk for next two years after enrolment, Children living with their biological mothers/parents, Families willing to sign a consent form.

Exclusion Criteria: History of illness involving calcium or bone metabolism, including stones of the urinary tract, Currently taking vitamin D supplements as treatment of any disease, Receiving immunosuppressive therapy (oral corticosteroids, chemotherapy) during the previous year, Known history of lactose intolerance or other contra-indications or a version to milk intake, Known hypercalcemia or hypercalciuria, Diabetes mellitus or past/current history of renal stones, and any known systemic, endocrine or metabolic disorder, Medications known to interact with vitamin D metabolism (steroids, thiazide diuretics, phenytoin, phenobarbitone, and antitubercular drugs), Hypersensitivity or allergy to any of the components used in nonfortified or fortified milk or oil, Any other reason which in the opinion of a Principal Investigator would interfere with the study shall be excluded.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals between the age 5 - 80 years will be enrolled.
Sampling Method: Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To assess impact on serum 25OHD concentrations | After December 2022
  Effect of consumption of fortified versus unfortified milk and oil on serum 25OHD concentrations of participants

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra B. Ghooi, Ph.D., Study Director — Scientia clinical services
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be shared by keeping names and other information of participant confidential.

REFERENCES:
- [Derived] Mandlik R, Deshpande S, Ladkat D, Patwardhan V, Khadilkar A. Impact of consumption of vitamin D fortified foods on serum vitamin D concentrations and vitamin D status in families living in Pune, India: an effectiveness study. Eur J Nutr. 2025 Mar 1;64(2):105. doi: 10.1007/s00394-025-03624-x. PMID 40025346